CLINICAL TRIAL: NCT02717923
Title: Maintenance Treatment With Capecitabine Plus Cetuximab After First-line 5-Fluorouracil-based Chemotherapy Plus Cetuximab for Patients With RAS Wild-type Metastatic Colorectal Cancer: a Single Arm, Open-label, Multi-center Clinical Trial
Brief Title: A Single Arm, Open-label Clinical Trial to Evaluate the Efficacy and Safety of Maintenance Treatment With Capecitabine Plus Cetuximab in Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: The First Affiliated Hospital of Nanchang University (Other); Hunan Cancer Hospital (Other); Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Xianglin Yuan, Professor, Chief physician, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJCC005
Record Dates: First submitted 2016-03-18; First posted 2016-03-24 (Estimated); Last update posted 2017-10-23 (Actual); Status verified 2017-10

CONDITIONS: Colorectal Neoplasms
Keywords: metastatic colorectal cancer; maintenance treatment; cetuximab
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine; Cetuximab

ARMS (1):
- Maintenance Treatment (Experimental): A single arm of maintenance treatment with capecitabine plus cetuximab after first-line 5-fluorouracil based standard chemotherapy plus cetuximab.
  Interventions: Other: maintenance treatment with capecitabine plus cetuximab

INTERVENTIONS:
Other: maintenance treatment with capecitabine plus cetuximab — Using a maintenance treatment strategy of capecitabine plus cetuximab as a treatment option in mCRC after first-line 5-FU-based chemotherapy plus cetuximab

SUMMARY:
This is a single arm, open-label, multi-center clinical trial to evaluate the efficacy and safety of maintenance treatment with capecitabine plus cetuximab after first-line 5-fluorouracil-based chemotherapy plus cetuximab for patients with RAS wild-type metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects has been fully understand this research and volunteered to sign the consent form;
2. Histologically and/or cytologically diagnosed with RAS wild-type metastatic metastatic colorectal cancer(Phase IIIc/IV), any other histological type is excluded;
3. Subjects with stable disease or better after induction treatment with eight to twelve 2-weekly cycles of 5FU-based standard chemotherapy;
4. ECOG Performance Status (ECOG PS) ≤1(0-1);
5. Evident measurable lesion(s) that meets the Response Evaluation Criteria in Solid Tumors (RECIST 1.1);
6. Expected survival>16 weeks.

Exclusion Criteria:

1. Subjects with presence of clinically detectable second primary malignant tumors at the enrollment, or other malignant tumors within the last 5 years (excluding adequately treated skin basal cell carcinoma or carcinoma in situ of cervix);
2. Clinical refractory diseases(including uncontrolled epilepsy),and affect survivor;
3. Central Nervous System (CNS) metastatic disease or prior cerebral metastasis;
4. Researchers think that the subjects exist any clinical or laboratory abnormalities or compliance issues and not suitable to participate in this clinical study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival of maintaining treatment（mPFS） | 5 years
  mPFS defined as time from randomisation to progression after maintenance

CONTACTS AND LOCATIONS:
Locations (1):
- Huazhong University of Science and Technology, Wuhan, Hubei, China

REFERENCES:
- [Background] Simkens LH, van Tinteren H, May A, ten Tije AJ, Creemers GJ, Loosveld OJ, de Jongh FE, Erdkamp FL, Erjavec Z, van der Torren AM, Tol J, Braun HJ, Nieboer P, van der Hoeven JJ, Haasjes JG, Jansen RL, Wals J, Cats A, Derleyn VA, Honkoop AH, Mol L, Punt CJ, Koopman M. Maintenance treatment with capecitabine and bevacizumab in metastatic colorectal cancer (CAIRO3): a phase 3 randomised controlled trial of the Dutch Colorectal Cancer Group. Lancet. 2015 May 9;385(9980):1843-52. doi: 10.1016/S0140-6736(14)62004-3. Epub 2015 Apr 7. PMID 25862517
- [Background] Hegewisch-Becker S, Graeven U, Lerchenmuller CA, Killing B, Depenbusch R, Steffens CC, Al-Batran SE, Lange T, Dietrich G, Stoehlmacher J, Tannapfel A, Reinacher-Schick A, Quidde J, Trarbach T, Hinke A, Schmoll HJ, Arnold D. Maintenance strategies after first-line oxaliplatin plus fluoropyrimidine plus bevacizumab for patients with metastatic colorectal cancer (AIO 0207): a randomised, non-inferiority, open-label, phase 3 trial. Lancet Oncol. 2015 Oct;16(13):1355-69. doi: 10.1016/S1470-2045(15)00042-X. Epub 2015 Sep 8. PMID 26361971
- [Derived] Wang L, Liu Y, Yin X, Fang W, Xiong J, Zhao B, Zhang M, Zou Y, Qiu H, Yuan X. Effect of Reduced-Dose Capecitabine Plus Cetuximab as Maintenance Therapy for RAS Wild-Type Metastatic Colorectal Cancer: A Phase 2 Clinical Trial. JAMA Netw Open. 2020 Jul 1;3(7):e2011036. doi: 10.1001/jamanetworkopen.2020.11036. PMID 32687588